CLINICAL TRIAL: NCT02734277
Title: Type 1 Diabetes Extension Study
Acronym: T1DES
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN066AI; NIAID CRMS ID#: 20722 (Other: DAIT NIAID)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitus; T1DM; T1D
Keywords: Insulin; Glucose Intolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood or urine tests as needed to follow-up on potential long term safety concerns with a particular therapeutic agent
  * Blood and urine samples for additional studies related to your diabetes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Detectable C-peptide by MMTT: Participants with detectable C-peptide at their:
  * Last Immune Tolerance Network (ITN) T1DM week 104 study visit,
  * Last AbATE (NCT00129259) follow-up visit, or
  * Last ITN066AI T1DES visit
  Detectable C-peptide is defined as a value above the lower limit of detection.
- Group 2:Undetectable C-peptide by MMTT: Participants without detectable C-peptide at their:
  * Last ITN T1DM week 104 study visit,
  * Last AbATE follow-up visit, or last
  * ITN066AI T1DES visit
  Undetectable C-peptide is defined as a value below the lower limit of detection.

SUMMARY:
This is a multi-center, prospective, non-interventional study that focuses on the long- term effects following participation in selected ITN new-onset Type1 Diabetes Mellitus studies with immunomodulatory agents (T1DM, T1D).

This observational study will:

* follow participants to determine how long they continue to produce insulin, and
* will also assess how changes in the immune system over time relate to the ability to produce insulin.

This information could help design better therapies for type 1 diabetes in the future.

DETAILED DESCRIPTION:
Depending upon a participant's level of insulin production, participation may be as short as one return visit or a maximum of five years. Evaluation visits will include:

* Overall health assessments
* Blood and urine collections
* Mixed meal tolerance test (MMTTs) for certain participants, per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Prior participant in an Immune Tolerance Network (ITN) executive committee approved T1DM study.
* Ability to sign informed consent/assent (as applicable for children).

Exclusion Criteria:

* Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial; or
* Inability to comply with the study visit schedule and required assessments.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Former participants in Immune Tolerance Network (ITN) new-onset Type 1 Diabetes Mellitus (T1DM) studies with immunomodulatory agents as the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2016-08-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Beta Cell Function by MMTT-Stimulated Mean C-peptide Area Under the Curve (AUC) | Baseline (Visit 0) to Month 60 (Year 5)
  Evaluation of changes in beta cell function over time will be measured by mixed-meal tolerance test (MMTT) -Stimulated mean C-Peptide area under the curve (AUC).
  C-peptide is released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin.
  Detectable C-peptide is defined as any value during a MMTT of ≥0.15 ng/mL.

SECONDARY OUTCOMES:
Change in Insulin Use in Units per Kilogram Body Weight Per Day | Baseline (Visit 0) to Month 60 (Year 5)
  The need to use exogenous insulin is an indication that the body is not producing enough endogenous insulin. Higher amounts of insulin use indicate higher disease activity.
Change in HbA1C | Baseline (Visit 0) to Month 60 (Year 5)
  Glycosylated hemoglobin (HbA1c) is a measure of the average plasma concentration of blood sugar (glucose) over the previous three months and measures the level of optimal management of underlying disease.
Count of Participant-Reported Major Hypoglycemic Events | Baseline (Visit 0) to Month 60 (Year 5)
  Major hypoglycemic events are defined as a glucose concentration <55 mg/dL (grades 2-5, NCI-CTCAE version 4.03), or clinically: involving seizure(s) or involving loss of consciousness (coma), or requiring assistance from another individual in order to recover.
Time to Undetectable C-Peptide | Baseline (Visit 0) to Month 60 (Year 5)
  To assess the longevity of beta cell function, time to undetectable C-peptide will be evaluated using Kaplan-Meier survival estimates.
Frequency of Grade 3 or Higher Adverse Events (AEs) of Interest | Baseline (Visit 0) to Month 60 (Year 5)
  Events of interest include but are not limited to:
  * Opportunistic and serious infections
  * Malignancy
  * Cardiovascular disease
  * Development of autoimmune disease(s)
  * Hypersensitivity reactions to unrelated allergens
  Reference for Grade 3 or higher AEs: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03 (June 14, 2010).
Severity of Grade 3 or Higher Adverse Events (AEs) of Interest | Baseline (Visit 0) to Month 60 (Year 5)
  Events of interest include but are not limited to:
  * Opportunistic and serious infections
  * Malignancy
  * Cardiovascular disease
  * Development of autoimmune disease(s)
  * Hypersensitivity reactions to unrelated allergens
  Reference for Grade 3 or higher AEs: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03 (June 14, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Linda A. DiMeglio, MD, MPH,MA, Study Chair — Riley Hospital for Children at Indiana University Health
Locations (12):
- United States (12):
  - UCSF School of Medicine, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado School of Medicine: Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Health Care Division of Pediatric Endocrinology, Iowa City, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Sanford Research, Sioux Falls, South Dakota
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in: 1.)ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools that are available to researchers who register online and subsequently receive DAIT approval; and 2.)TrialShare, a clinical trials research portal developed by the Immune Tolerance Network that makes data from the consortium's clinical trials publicly available without charge.
Time Frame: After completion of the study.
Access Criteria: Will be available to the public.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- [Background] Herold KC, Gitelman SE, Ehlers MR, Gottlieb PA, Greenbaum CJ, Hagopian W, Boyle KD, Keyes-Elstein L, Aggarwal S, Phippard D, Sayre PH, McNamara J, Bluestone JA; AbATE Study Team. Teplizumab (anti-CD3 mAb) treatment preserves C-peptide responses in patients with new-onset type 1 diabetes in a randomized controlled trial: metabolic and immunologic features at baseline identify a subgroup of responders. Diabetes. 2013 Nov;62(11):3766-74. doi: 10.2337/db13-0345. Epub 2013 Jul 8. PMID 23835333
- [Background] Rigby MR, Harris KM, Pinckney A, DiMeglio LA, Rendell MS, Felner EI, Dostou JM, Gitelman SE, Griffin KJ, Tsalikian E, Gottlieb PA, Greenbaum CJ, Sherry NA, Moore WV, Monzavi R, Willi SM, Raskin P, Keyes-Elstein L, Long SA, Kanaparthi S, Lim N, Phippard D, Soppe CL, Fitzgibbon ML, McNamara J, Nepom GT, Ehlers MR. Alefacept provides sustained clinical and immunological effects in new-onset type 1 diabetes patients. J Clin Invest. 2015 Aug 3;125(8):3285-96. doi: 10.1172/JCI81722. Epub 2015 Jul 20. PMID 26193635
- [Background] Rigby MR, DiMeglio LA, Rendell MS, Felner EI, Dostou JM, Gitelman SE, Patel CM, Griffin KJ, Tsalikian E, Gottlieb PA, Greenbaum CJ, Sherry NA, Moore WV, Monzavi R, Willi SM, Raskin P, Moran A, Russell WE, Pinckney A, Keyes-Elstein L, Howell M, Aggarwal S, Lim N, Phippard D, Nepom GT, McNamara J, Ehlers MR; T1DAL Study Team. Targeting of memory T cells with alefacept in new-onset type 1 diabetes (T1DAL study): 12 month results of a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):284-94. doi: 10.1016/S2213-8587(13)70111-6. Epub 2013 Sep 23. PMID 24622414
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait